CLINICAL TRIAL: NCT03991169
Title: Pilot Pragmatic Clinical Trial of Oral Iron Therapy in Children With Chronic Kidney Disease
Brief Title: Oral Iron in Children With Chronic Kidney Disease
Acronym: FeTCh-CKD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1812019836
Record Dates: First submitted 2019-06-06; First posted 2019-06-19 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Chronic Kidney Insufficiency; Chronic Kidney Diseases
Keywords: Anemia; Iron; Children; Chronic kidney disease (CKD); Appetite; Physical activity; Muscle strength
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia; Motor Activity | interventions — ferrous sulfate; Iron-Dextran Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oral Iron therapy (Experimental): Participant will receive oral iron therapy.
  Interventions: Drug: Ferrous Sulfate
- No oral iron therapy (No Intervention): Participant will not receive oral iron therapy for 3 months.

INTERVENTIONS:
Drug: Ferrous Sulfate — Oral iron will be given in the form of immediate-release iron sulfate, 3-6 mg/kg/day of elemental iron to children with body weight ≤43 kg, and 65 mg of elemental iron (325 mg of iron sulfate) to children with body weight >43 kg.
  Other Names: iron sulfate
  Arms: Oral Iron therapy

SUMMARY:
This is a pilot clinical trial of oral iron therapy in children with chronic kidney disease (CKD) and mild anemia. Eligible children will be randomized into a standard of care (iron sulfate) arm vs. no iron therapy arm for 3 months. The outcomes will include muscle strength, physical activity, and changes in eating behavior, which will be measured at enrollment and at the end of the study period.

ELIGIBILITY:
Key inclusion criteria:

* Age 1-21 years old (muscle strength will be assessed only in children >3 year old)
* Estimated glomerular filtration rate (GFR) < 90 ml/min/1.73m2 by bedside Schwartz formula [height (cm) *0.413 / serum creatinine (mg/dL)]
* Hemoglobin (Hb) more or equal than 9.0 at the previous clinic visit
* Hb less than 11.5 g/dL in children younger than 5 years Hb less than 12.0 g/dL in children 5-12 years Hb <12.5 g/dL in children 12-15 yrs and females >15 yrs. Hb <13.5 g/dL in males >15 years (all at the previous clinic visit)

Children with transferrin saturation ≤ 20% AND serum ferritin ≤ 100 ng/mL will be randomized into one of the arms

Key exclusion criteria:

* Transferrin saturation <5%
* Serum ferritin < 10 ng/mL
* Iron therapy or erythrocyte stimulating agents (erythropoietin) therapy within 3 months prior to randomization
* Blood transfusion within 4 months prior to enrollment
* Children on hemodialysis
* Rapidly deteriorating kidney function or expectation for transplantation or dialysis in less than 3 months
* Pregnancy and breast-feeding

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-04-19 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in muscle strength | 0 and 3 months
  Hand-grip strength measured by a dynamometer
Change in the percentage of transferrin saturation in the participants' blood | 0 and 3 months
  Transferrin saturation is a medical laboratory value, measured as a percentage. It is the value of serum iron concentration divided by the total iron-binding capacity. For instance, a value of 15% means that 15% of iron-binding sites of transferrin are being occupied by iron.
  Blood will be collected with the venopuncture used for clinically indicated blood tests at routine clinic visits

SECONDARY OUTCOMES:
Change in sedentary time | 0 and 3 months
  Sedentary time (in minutes per day) will be measured by actigraphy. Actigraph is a monitor that looks like a wristband or a watch that measures and records body movements throughout the day. Participating children will wear actigraphs for 7 days in the beginning and 7 days at the conclusion of the study.
Change in the percent of skeletal muscle mass | 0 and 3 months
  Percent of skeletal muscle mass out of body weight will be measured using bio-electrical impedance analysis.
Change in eating behavior | 0 and 3 months
  Appetite / eating behavior assessed using Children's Eating Behavior Questionnaire (CEBQ). It is a parent-report measure comprised of 35 items, each rated as "Never", "Rarely", "Sometimes", "Often", "Always". The answers will be grouped into the domains to assess eating styles of the participating children, such as: "Enjoyment of food", "Slowness in eating", "Emotional under-eating", "Food fussiness".
Change in quality of life: PROMIS | 0 and 3 months
  Quality of life will be assessed in the Fatigue, and Physical Activity domains using the Patient-Reported Outcomes Measurement Information System (PROMIS), developed by the National Institutes of Health. PROMIS measures use a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
  Higher scores will mean more Fatigue and more Physical Activity respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Oleh Akchurin, M.D., Principal Investigator — Weill Cornell College of Medicine
Locations (2):
- United States (2):
  - Weill Cornell Medicine / New York Presbyterian Hospital, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No